CLINICAL TRIAL: NCT04474639
Title: Diastolic Dysfunction Assessment of the Left Ventricle Using Spectral Analysis of a Single Lead ECG
Brief Title: Determination of Diastolic Dysfunction by Single Lead Electrocardiogram
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 1305
Record Dates: First submitted 2020-06-22; First posted 2020-07-17 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Diastolic Function
Keywords: diastolic function; heart failure; spectral analysis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with diastolic dysfunction: patients with diastolic dysfunction of the left ventricle confirmed by the results of the echocardiography (septal e' >=8, and lateral e'>=10 and left atrium <34 ml/m2) and by results of the spectral analysis of electrocardiogram (the parameters listed below will be calculated as the median of the tact-cycle: TpTe, VAT, QTc, QT / TQ, QRS_E, T_E, TP_E, BETA, BETA_S, BAD_T, QRS_D1_ons, QRS_D1_offs, QRS_D2, QRS_Ei (i = 1,2,3,4), T_Ei (i= 1,2,3,4), HFQRS, QRSw, RA, SA, TA).
  Interventions: Device: echocardiographic examination
- without diastolic dysfunction: patients without diastolic dysfunction of the left ventricle confirmed by the results of the echocardiography (septal e'<8, and lateral e'<10 and left atrium >=34 ml/m2) and by results of the spectral analysis of electrocardiogram (the parameters listed below will be calculated as the median of the tact-cycle: TpTe, VAT, QTc, QT / TQ, QRS_E, T_E, TP_E, BETA, BETA_S, BAD_T, QRS_D1_ons, QRS_D1_offs, QRS_D2, QRS_Ei (i = 1,2,3,4), T_Ei (i= 1,2,3,4), HFQRS, QRSw, RA, SA, TA).
  Interventions: Device: echocardiographic examination

INTERVENTIONS:
Device: echocardiographic examination — conducting an echocardiographic study according to a standard protocol with the determination of diastolic dysfunction of the left ventricle

SUMMARY:
It is a prospective, controlled, single-center, non-randomized, observational study.

From September 2019 to December 2020, the study plans to prospectively include 400 patients aged 18 to 90 years.

Every patients will undergo an echocardiographic examination with assessment diastolic dysfunction of the left ventricle, and registration of an electrocardiogram using a single lead ECG monitor CardioQvark (in I standard lead) for 3 minutes. All patients will be divided into 2 main groups: with diastolic dysfunction of the left ventricle, confirmed by the results of the echocardiography and without. A spectral analysis of the electrocardiogram will be performed using a continuous wavelet transform.

The result of this study will be the identification of ECG parameters that will correlate with LV diastolic dysfunction.

DETAILED DESCRIPTION:
It is a prospective, controlled, single-center, non-randomized, observational study.

From September 2019 to December 2020, the study plans to prospectively include 400 patients aged 18 to 90 years.

The goal of study is reveal single parameters of the electrocardiogram, which a good correlation with left ventricular diastolic dysfunction (LV DD), discovered during echocardiography.

Investigators plan to assess the diagnostic effectiveness of the spectral analysis of electrocardiograms obtained using a single-lead portable ECG monitor.

All subjects will undergo an echocardiographic examination of the heart with a determination of diastolic dysfunction of the left ventricle and will be divided into 2 main groups: with diastolic dysfunction of the left ventricle, confirmed by the results of the echocardiography and without.

At the same time, for all patients single-lead ECG will be recorded (in turn of leads I) for 3 minutes with further spectral analysis of the data obtained.

A single-lead ECG monitor CardioQvark is designed as an iPhone cover. It is registered with the Federal Service for Health Supervision on February 15, 2019. RZN No. 2019/8124.

Then a spectral analysis of the electrocardiogram will be performed using a continuous wavelet transform, the principles of which are based on the Fourier transform.

The analysis implies an assessment of the following parameters (the parameters listed below will be calculated as the median of the tact-cycle):

* TpTe - time from peak to end of the T-wave
* VAT - time from the beginning of the QRS to the R-peak
* QTc - corrected QT interval.
* QT / TQ - the ratio of QT length to TQ length (from the end of T to the beginning of the QRS of the next complex).
* QRS_E - the total energy of the QRS wave based on the wavelet transform
* T_E - T-wave total energy based on wavelet transform
* TP_E- energy of the main tooth of the T-wave based on the wavelet transform
* BETA, BETA_S - T-wave asymmetry coefficients (simple and smooth versions)
* BAD_T - flag of T-wave quality (whether expressed in the current lead
* QRS_D1_ons - energy of the leading edge of the R-wave (based on the "first derivative" wavelet transform)
* QRS_D1_offs - energy of the trailing edge of the R-wave (based on the "first derivative" wavelet transform)
* QRS_D2 - peak energy of the R-wave (based on the "second derivative" wavelet transform)
* QRS_Ei (i = 1,2,3,4) - QRS-wave energy in 4 frequency ranges (2-4-8-16-32 Hz) based on wavelet transform
* T_Ei (i = 1,2,3,4) - T-wave energy in 4 frequency ranges (2-4-6-8-10 Hz) based on wavelet transform
* HFQRS - the amplitude of the RF components of the QRS wave

Additionally used parameters:

* TpTe, VAT, QTc - are duplicated to control the correctness of the record processing (the value of the UCC should be approximately equal to the median of the tick-by-bar).
* QRSw - QRS width.
* RA, SA, TA - the amplitudes of the R, S, T-waves, respectively, are used to normalize the parameters listed above.

Statistical processing of results: SPSS Statistics Version 26 is a computer program for statistical processing of data.

The result of this study will be the identification of ECG parameters that will correlate with LV diastolic dysfunction, and by which it will be possible to determine its presence and degree in the future.

Investigators also plan to analyze ECG parameters characteristic of patients with LV diastolic dysfunction in different population groups:

* patients suffering from high blood pressure with patients without the above pathology
* patients with zones of a- and hypokinesis according to echocardiography as a result of a coronary circulation disorder
* patients suffering from atrial fibrillation with patients without this pathology
* men / women
* patients of different age groups

During statistical processing of the data, the following will be calculated: sensitivity, specificity, prognostic value of positive and negative results, likelihood ratio, area under ROC - curve, correlation coefficient. it is planned to obtain data on the diagnostic effectiveness of the proposed approach, as well as on individual parameters of the electrocardiogram in the diagnosis of diastolic dysfunction of the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* The presence of written informed consent of the patient to participate in the study
* Age from 18 years to 90 years
* Outpatient treatment and / or hospitalization in a research center

Exclusion Criteria:

* Reluctance of the patient to participate in the study
* Poor quality ECG recording on a single-channel ECG monitor
* Poor visualization of the heart during echocardiographic study
* Acute psychotic reactions that arose during research
* An exacerbation of chronic diseases requiring treatment tactics for the patient and preventing his further participation in the study.

Non-inclusion criteria:

* The presence of conduction disturbances in patients that impede ECG analysis (WPW syndrome, sinoatrial block of degrees 2 and 3, atrioventricular block 3 degrees, complete block of the left bundle branch block, complete block of the right bundle branch block)
* Conditions that can impair ECG recording quality (Parkinson's disease, essential tremor)
* The inability to assess diastolic function during echocardiography
* Mental illness
* Diseases with an expected life expectancy of less than 2 years
* Patients with diffuse hypokinesis of the left ventricle with a reduced ejection fraction (less than 30%)
* Patients with a pacemaker installed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients aged 18 to 90 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
determination of sensitivity of LV DD using a single-channel ECG monitor CardioQvark | through study completion, an average of 2 years
  comparison of the presence of LV DD detected by the results of an echocardiographic study with the results of the presence of LV DD obtained using the mathematical model of a single-channel ECG of the CardioQvark monitor
determination of specificity of LV DD using a single-channel ECG monitor CardioQvark | through study completion, an average of 2 years
  comparison of the presence of LV DD detected by the results of an echocardiographic study with the results of the presence of LV DD obtained using the mathematical model of a single-channel ECG of the CardioQvark monitor
determination of prognostic value of positive and negative results of LV DD using a single-channel ECG monitor CardioQvark | through study completion, an average of 2 years
  comparison of the presence of LV DD detected by the results of an echocardiographic study with the results of the presence of LV DD obtained using the mathematical model of a single-channel ECG of the CardioQvark monitor
determination of likelihood ratio of LV DD using a single-channel ECG monitor CardioQvark | through study completion, an average of 2 years
  comparison of the presence of LV DD detected by the results of an echocardiographic study with the results of the presence of LV DD obtained using the mathematical model of a single-channel ECG of the CardioQvark monitor
determination of area under ROC - curve of LV DD using a single-channel ECG monitor CardioQvark | through study completion, an average of 2 years
  comparison of the presence of LV DD detected by the results of an echocardiographic study with the results of the presence of LV DD obtained using the mathematical model of a single-channel ECG of the CardioQvark monitor
determination of correlation coefficient of LV DD using a single-channel ECG monitor CardioQvark | through study completion, an average of 2 years
  comparison of the presence of LV DD detected by the results of an echocardiographic study with the results of the presence of LV DD obtained using the mathematical model of a single-channel ECG of the CardioQvark monitor

SECONDARY OUTCOMES:
significance of the parameter TpTe on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter VAT on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QTc on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QT / TQ on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_E on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter T_E on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter TP_E on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter BETA on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter BETA_S on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter BAD_T on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_D1_ons on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_D1_offs on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_D2 on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_Ei on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter T_Ei on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter HFQRS on the ECG in the determination of LV DD | through study completion, an average of 2 years
  an ECG spectral analysis will be performed using the Fourier Transform

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kopylov, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University); Natalia Kuznetsova, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
It is not possible to provide documentation due to the prohibition received from the local ethics committee